CLINICAL TRIAL: NCT03240926
Title: Loop Band Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spry Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 32315
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: COPD
Keywords: COPD; COPD Exacerbation; COPD Asthma; COPD Bronchitis; COPD, Severe Early-Onset
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Disease, Chronic Obstructive, Severe Early-Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Loop Band (Experimental): Measure accuracy of vital sign measurements
  Interventions: Device: Loop Band

INTERVENTIONS:
Device: Loop Band — Application of Loop band on radial artery of the opposite wrist that the Anesthesiologist has placed the Arterial line.

SUMMARY:
The main purpose of this study is to assess the accuracy of a non-invasive wearable technology in the form of a wristband.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the accuracy of a non-invasive wearable technology in the form of a wristband. This wristband (Loop Band) uses optical sensors and spectrometry to measure and estimate vitals as well as a full blood gas panel; comparable to the standard method of an invasive arterial line and pressure transducer. The investigators aim to show equivalence of clinical physiologic outcome measurements with the Loop Band relative to current methods (i.e. arterial lines, etc.). In addition, this study aims to validate this wearable technology as a potential alternative to invasive measurements, to reduce complications, and improve accuracy in regards to patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient has capacity to consent for the study.
* Anesthetic plan for an arterial line for vital sign monitoring during their surgical procedure.

Exclusion Criteria:

* Active Atrial Fibrillation
* Active C-difficile
* Amputation of the arm at the wrist or above
* The Investigator and/or Clinical Research Nurse will conduct a visual inspection for attributes that may diminish device accuracy. These include but are not limited to: tattoos over the radial artery, burns or heavy scarring over the radial artery, fragile skin, any skin diseases affecting the wrist or arm, Physician discretion-any condition deemed inappropriate that will preclude use of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Device Equivalence in clinical outcome measures (heart rate, blood oxygenation, carboxyhemoglobin level, end tidal carbon dioxide, and respiratory rate) measured by Arterial Line. | intraoperative
  Equivalence in clinical outcome measures (heart rate, blood oxygenation, carboxyhemoglobin level, end tidal carbon dioxide, and respiratory rate etc.) with the Loop Band relative to current methods (i.e. arterial lines, etc.) during a surgical procedure.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | intraoperative
  Evaluate safety data based on reported Adverse Events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Harry Bowles, MD, Principal Investigator — Spry Health
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No